CLINICAL TRIAL: NCT01326403
Title: Tranexamic Acid in Hip Fracture Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Michal Roll PhD,MBA (Other Government)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor-Investigator, Michal Roll PhD,MBA, division of research and development TASMC, Tel-Aviv Sourasky Medical Center
Organization: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: TASMC-11-ES-0129-CTIL
Record Dates: First submitted 2011-03-21; First posted 2011-03-30 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: Closed Fracture of Hip
Keywords: proximal; hip; fractures
MeSH Terms: conditions — Fractures, Bone | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Patients will receive IV Tranexamic acid 1 gram upon diagnosis and consent in the emergency room. A second 1 gram in a slow drip during the next 8 hours.
  Interventions: Drug: Tranexamic acid
- GROUP B (Experimental): Patients will receive IV Tranexamic acid 1 gram five minutes before skin incision and a second 1 gram in a slow drip during the next 8 hours.
  Interventions: Drug: Tranexamic acid
- GROUP C (Placebo Comparator): A control group will only receive placebo in the emergency room and in the OR.
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — GROUP A - receive IV Tranexamic acid 1 gram upon diagnosis and consent in the emergency room. A second 1 gram in a slow drip during the next 8 hours.
  GROUP B - IV Tranexamic acid 1 gram five minutes before skin incision and a second 1 gram in a slow drip during the next 8 hours.
  Group C - A control group will only receive placebo in the emergency room and in the OR.
  Other Names: placebo group; post injury group; preoperative group

SUMMARY:
This is a randomized controlled trial comparing the use of tranexamic acid to placebo in patients admitted to hospital with a hip fracture.

DETAILED DESCRIPTION:
1. transfusion of allogeneic RBC's is not free of adverse events and has been associated with an increased risk of postoperative infection
2. Tranexamic acid in trauma patients has been shown to reduce 30-day mortality. Hospital trauma protocol includes tranexamic acid in patients with major bleeding.
3. Tranexamic acid in orthopedic elective joint reconstruction surgery has been shown to substantially decrease bleeding in knee and hip arthroplasty.
4. in hip fracture surgery, transexamic acid reduces erythrocyte transfusion rate but may promote a hypercoagulable state.
5. Tranexamic acid is an antifibrinolytic drug that inhibits plasminogen from turning into plasmin thereby inhibiting clot breakdown.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency room with proximal hip fractures (31A-31B according to the Muller AO classification of fractures - long bones).
* Patients mentally capable of giving informed consent.

Exclusion Criteria:

1. Vascular events within the last 2 months such as CVA, TIA, ACS, MI, DVT or arterial thrombosis.
2. Patients receiving anticoagulation therapy with Coumadin or Plavix.
3. Pregnancy and breastfeeding females.
4. Previous arterial or venous thrombosis
5. History of seizures.
6. Creatinine >2.
7. Oestroprogestive therapy.
8. Multiple fractures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Total amount of blood loss per patient from admission to day 5 post-op | 5 DAYS

SECONDARY OUTCOMES:
Number of packed cell transfusion per patient. | 5 DAYS
Initial functional outcome and feeling of well-being. | 5 days
thromboembolic events | 5 days
post-operative bacterial infection | 5 days
30 day mortality rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: ELI SHTEINBERG, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel